CLINICAL TRIAL: NCT02570425
Title: THE HCP ELIOT STUDY: Comparing Maintenance of Device Mastery With TURBOHALER© vs. SPIROMAX© in Healthcare Professionals naïve to Both Devices (The Easy Low Instruction Over Time [ELIOT] Study)
Brief Title: Comparing Maintenance of Device Mastery With Turbohaler© vs. Spiromax© in Healthcare Professionals naïve to Both Devices
Acronym: HCP-ELIOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Teva Branded Pharmaceutical Products R&D, Inc. (Industry); University of Sydney (Other); Woolcock Institute of Medical Research (Other); University of Technology, Sydney (Other); The University of New South Wales (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: OR00114
Record Dates: First submitted 2015-08-07; First posted 2015-10-07 (Estimated); Results first posted 2016-05-30 (Estimated); Last update posted 2016-05-30 (Estimated); Status verified 2016-04

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spiromax followed by Turbohaler (Placebo Comparator): Training on BF Spiromax followed by SYMBICORT Turbohaler
  Interventions: Device: Training on BF Spiromax followed by SYMBICORT Turbohaler; Device: Training on SYMBICORT Turbohaler followed by BF Spiromax
- Turbohaler followed by Spiromax (Placebo Comparator): Training on SYMBICORT Turbohaler followed by BF Spiromax
  Interventions: Device: Training on BF Spiromax followed by SYMBICORT Turbohaler; Device: Training on SYMBICORT Turbohaler followed by BF Spiromax

INTERVENTIONS:
Device: Training on BF Spiromax followed by SYMBICORT Turbohaler — Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
Device: Training on SYMBICORT Turbohaler followed by BF Spiromax — Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.

SUMMARY:
This study is conducted to assess the ease of device mastery of a placebo SYMBICORT TURBOHALER vs a placebo Budesonide/Formoterol SPIROMAX device among healthcare professionals in-training (HCP).

DETAILED DESCRIPTION:
The purpose of this study is to identify how intuitive devices are to use and what level of training is required to ensure that HCPs are able to demonstrate the correct technique. The two devices examined will be the SYMBICORT TURBOHALER and placebo Budesonide/Formoterol SPIROMAX device among healthcare professionals (HCP).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent is obtained and dated by the participant before conducting any study related procedures.
* The participant is a student that is currently enrolled in the University where the study is conducted
* The participant must be willing and able to comply with study restrictions and to remain at the study site for the required duration during the study period, and willing to return to the site for the follow up evaluation as specified in this protocol.
* The participant has not previously used or received training in the use of either the SPIROMAX or the TURBOHALER in the last 6 months

Exclusion Criteria:

* Participants will be excluded from participating in this study if they have asthma.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 516 (Actual)
Dates: Start 2014-07; Primary Completion 2014-09 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sinthia Bosnic-Anticevich, PhD, Principal Investigator — University of Sydney

IPD SHARING:
Plan to Share IPD: Undecided
Decision has not been made

REFERENCES:
- [Background] Al-Jahdali H, Ahmed A, Al-Harbi A, Khan M, Baharoon S, Bin Salih S, Halwani R, Al-Muhsen S. Improper inhaler technique is associated with poor asthma control and frequent emergency department visits. Allergy Asthma Clin Immunol. 2013 Mar 6;9(1):8. doi: 10.1186/1710-1492-9-8. PMID 23510684
- [Background] Basheti IA, Armour CL, Reddel HK, Bosnic-Anticevich SZ. Long-term maintenance of pharmacists' inhaler technique demonstration skills. Am J Pharm Educ. 2009 Apr 7;73(2):32. doi: 10.5688/aj730232. PMID 19513170
- [Background] Basheti IA, Armour CL, Bosnic-Anticevich SZ, Reddel HK. Evaluation of a novel educational strategy, including inhaler-based reminder labels, to improve asthma inhaler technique. Patient Educ Couns. 2008 Jul;72(1):26-33. doi: 10.1016/j.pec.2008.01.014. Epub 2008 Mar 7. PMID 18314294
- [Background] Beasley R, Crane J, Lai CK, Pearce N. Prevalence and etiology of asthma. J Allergy Clin Immunol. 2000 Feb;105(2 Pt 2):S466-72. doi: 10.1016/s0091-6749(00)90044-7. PMID 10669525
- [Background] Cain WT, Cable G, Oppenheimer JJ. The ability of the community pharmacist to learn the proper actuation techniques of inhaler devices. J Allergy Clin Immunol. 2001 Dec;108(6):918-20. doi: 10.1067/mai.2001.119153. PMID 11742268
- [Background] National Asthma Education and Prevention Program. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol. 2007 Nov;120(5 Suppl):S94-138. doi: 10.1016/j.jaci.2007.09.043. PMID 17983880
- [Background] Giraud V, Roche N. Misuse of corticosteroid metered-dose inhaler is associated with decreased asthma stability. Eur Respir J. 2002 Feb;19(2):246-51. doi: 10.1183/09031936.02.00218402. PMID 11866004
- [Background] Gupta R, Sheikh A, Strachan DP, Anderson HR. Burden of allergic disease in the UK: secondary analyses of national databases. Clin Exp Allergy. 2004 Apr;34(4):520-6. doi: 10.1111/j.1365-2222.2004.1935.x. PMID 15080802
- [Background] Hanania NA, Wittman R, Kesten S, Chapman KR. Medical personnel's knowledge of and ability to use inhaling devices. Metered-dose inhalers, spacing chambers, and breath-actuated dry powder inhalers. Chest. 1994 Jan;105(1):111-6. doi: 10.1378/chest.105.1.111. PMID 8275720
- [Background] Haughney J, Price D, Barnes NC, Virchow JC, Roche N, Chrystyn H. Choosing inhaler devices for people with asthma: current knowledge and outstanding research needs. Respir Med. 2010 Sep;104(9):1237-45. doi: 10.1016/j.rmed.2010.04.012. Epub 2010 May 15. PMID 20472415
- [Background] Haughney J, Price D, Kaplan A, Chrystyn H, Horne R, May N, Moffat M, Versnel J, Shanahan ER, Hillyer EV, Tunsater A, Bjermer L. Achieving asthma control in practice: understanding the reasons for poor control. Respir Med. 2008 Dec;102(12):1681-93. doi: 10.1016/j.rmed.2008.08.003. Epub 2008 Sep 23. PMID 18815019
- [Background] Ovchinikova L, Smith L, Bosnic-Anticevich S. Inhaler technique maintenance: gaining an understanding from the patient's perspective. J Asthma. 2011 Aug;48(6):616-24. doi: 10.3109/02770903.2011.580032. Epub 2011 May 31. PMID 21623690
- [Background] Papi A, Haughney J, Virchow JC, Roche N, Palkonen S, Price D. Inhaler devices for asthma: a call for action in a neglected field. Eur Respir J. 2011 May;37(5):982-5. doi: 10.1183/09031936.00150910. No abstract available. PMID 21532013
- [Background] Pinnock H, Thomas M, Tsiligianni I, Lisspers K, Ostrem A, Stallberg B, Yusuf O, Ryan D, Buffels J, Cals JW, Chavannes NH, Henrichsen SH, Langhammer A, Latysheva E, Lionis C, Litt J, van der Molen T, Zwar N, Williams S. The International Primary Care Respiratory Group (IPCRG) Research Needs Statement 2010. Prim Care Respir J. 2010 Jun;19 Suppl 1(Suppl 1):S1-20. doi: 10.4104/pcrj.2010.00021. PMID 20514388
- [Background] Inhaler Error Steering Committee; Price D, Bosnic-Anticevich S, Briggs A, Chrystyn H, Rand C, Scheuch G, Bousquet J. Inhaler competence in asthma: common errors, barriers to use and recommended solutions. Respir Med. 2013 Jan;107(1):37-46. doi: 10.1016/j.rmed.2012.09.017. Epub 2012 Oct 23. PMID 23098685
- [Derived] Price DB, Thomas V, Richard Dekhuijzen PN, Bosnic-Anticevich S, Roche N, Lavorini F, Raju P, Freeman D, Nicholls C, Small IR, Sims E, Safioti G, Canvin J, Chrystyn H. Evaluation of inhaler technique and achievement and maintenance of mastery of budesonide/formoterol Spiromax(R) compared with budesonide/formoterol Turbuhaler(R) in adult patients with asthma: the Easy Low Instruction Over Time (ELIOT) study. BMC Pulm Med. 2018 Jun 28;18(1):107. doi: 10.1186/s12890-018-0665-x. PMID 29954359

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants were re-randomised to either the BF Spiromax first or Symbicort Turbohaler first at each visit.
Groups:
- Placebo Comparator: Spiromax Followed by Turbohaler: Training on BF Spiromax followed by SYMBICORT Turbohaler
- Placebo Comparator: Turbohaler Followed by Spiromax: Training on SYMBICORT Turbohaler followed by BF Spiromax
Period: Visit 1
Arm/Group | Placebo Comparator: Spiromax Followed by Turbohaler | Placebo Comparator: Turbohaler Followed by Spiromax
Started | 274 | 242
Completed | 274 | 242
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | Placebo Comparator: Spiromax Followed by Turbohaler | Placebo Comparator: Turbohaler Followed by Spiromax
Started | 251 (In total 18 patients who completed Visit 1, did not attend Visit 2.) | 247 (In total 18 patients who completed Visit 1, did not attend Visit 2.)
Completed | 251 | 247
Not Completed | 0 | 0
Period: Visit 3
Arm/Group | Placebo Comparator: Spiromax Followed by Turbohaler | Placebo Comparator: Turbohaler Followed by Spiromax
Started | 229 (In total 38 patients who completed Visit 2, did not attend Visit 3.) | 231 (In total 38 patients who completed Visit 2, did not attend Visit 3.)
Completed | 229 | 231
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SYMBICORT Turbohaler® First, Then Spiromax®: Training HCPs with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: Budesonide/Formoterol (BF) Spiromax®: Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: SYMBICORT® Turbohaler: Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Training HCPs: Training HCPS with both devices using a 6-level system to examine the number of levels required to acquire mastery of device at baseline
- Budesonide/Formoterol (BF) Spiromax® First, Then Turbohaler®: Traing HCPs with a placebo comparator: Budesonide/Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: Budesonide/Formoterol (BF) Spiromax®: Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: SYMBICORT® Turbohaler: Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Training HCPs: Training HCPS with both devices using a 6-level system to examine the number of levels required to acquire mastery of device
- Total: Total of all reporting groups
Arm/Group | SYMBICORT Turbohaler® First, Then Spiromax® | Budesonide/Formoterol (BF) Spiromax® First, Then Turbohaler® | Total
Number analyzed (Participants) | 242 | 274 | 516
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 242 | 274 | 516
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.9 (4.5) | 22.3 (4.7) | 22.6 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 146 | 169 | 315
  Male | 96 | 105 | 201
Region of Enrollment [Number; unit: participants]
  Australia | 242 | 274 | 516

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Maintaining Correct Inhaler Technique for Spiromax Compared With Turbohaler 4 Weeks After Training as Assessed by Expert Assessor
Description: Examine if recall of device mastery is superior for the SPIROMAX inhaler as compared to the TURBOHALER after training to device mastery on both devices.
  The proportion of subjects achieving mastery of inhaler technique between the two inhaler devices was compared using McNemar's test of equality of paired proportions with a 0.050 two- sided significance level. A Conditional Logistic Regression Model was used to quantify the difference between the two inhalers by calculating the odds ratio for achieving mastery for Spiromax® (with Turbohaler® as the reference device) along with a 95% confidence interval for quantifying the precision of the odds ratio estimate.
Time Frame: 4 weeks
Measure: Number; unit: percent of participants
Groups:
- SYMBICORT Turbohaler®: Training HCPs with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: Budesonide/Formoterol (BF) Spiromax®: Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: SYMBICORT® Turbohaler: Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Training HCPs: Training HCPS with both devices using a 6-level system to examine the number of levels required to acquire mastery of device at baseline
- Budesonide/Formoterol (BF) Spiromax®: Traing HCPs with a placebo comparator: Budesonide/Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: Budesonide/Formoterol (BF) Spiromax®: Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: SYMBICORT® Turbohaler: Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Training HCPs: Training HCPS with both devices using a 6-level system to examine the number of levels required to acquire mastery of device
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 498 | 498
percent of participants | 40 | 64

2. Secondary Outcome: Percentage of Participants Achieving Device Mastery at the End of Level 1 Out of a 6 Level Training Process as Assessed by Expert Assessor
Description: Examined for both at the end of level 1 (out of 6 level training process). This will be compared using McNemar's test of equality of paired proportions with a 0.050 two- sided significance level. A Conditional Logistic Regression Model was used to quantify the difference between the two inhalers by calculating the odds ratio for achieving mastery for Spiromax® (with Turbohaler® as the reference device) along with a 95% confidence interval for quantifying the precision of the odds ratio estimate.
Time Frame: 0 weeks (Visit 1)
Measure: Number; unit: percent of participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 516 | 516
percent of participants | 4 | 22

3. Secondary Outcome: Percentage of Participants Achieving Device Mastery at the End of Level 2 Out of a 6 Level Training Process as Assessed by Expert Assessor
Description: Examined for both at the end of level 2 (out of 6 level training process). This will be compared using McNemar's test of equality of paired proportions with a 0.050 two- sided significance level. A Conditional Logistic Regression Model was used to quantify the difference between the two inhalers by calculating the odds ratio for achieving mastery for Spiromax® (with Turbohaler® as the reference device) along with a 95% confidence interval for quantifying the precision of the odds ratio estimate.
Time Frame: 0 weeks (Visit 1)
Measure: Number; unit: percent of participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 516 | 516
percent of participants | 31 | 58

4. Secondary Outcome: Percentage of Participants Achieving Device Mastery at the End of Level 1 Out of a 6 Level Training Process at Week 4 as Assessed by Expert Assessor
Description: Examined at the end of level 1 (out of 6 level training process). This will be compared using McNemar's test of equality of paired proportions with a 0.050 two- sided significance level. A Conditional Logistic Regression Model was used to quantify the difference between the two inhalers by calculating the odds ratio for achieving mastery for Spiromax® (with Turbohaler® as the reference device) along with a 95% confidence interval for quantifying the precision of the odds ratio estimate.
Time Frame: 4 weeks
Measure: Number; unit: percent of participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 498 | 498
percent of participants | 40 | 64

5. Secondary Outcome: Percentage of Participants Achieving Device Mastery at the End of Level 2 Out of a 6 Level Training Process at Week 4 as Assessed by Expert Assessor
Description: Examined at the end of level 2 (out of 6 level training process). This will be compared using McNemar's test of equality of paired proportions with a 0.050 two- sided significance level. A Conditional Logistic Regression Model was used to quantify the difference between the two inhalers by calculating the odds ratio for achieving mastery for Spiromax® (with Turbohaler® as the reference device) along with a 95% confidence interval for quantifying the precision of the odds ratio estimate.
Time Frame: 4 weeks
Measure: Number; unit: percent of participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 498 | 498
percent of participants | 77 | 86

6. Secondary Outcome: Percentage of Participants Achieving Device Mastery at the End of Level 1 Out of a 6 Level Training Process at Week 8 as Assessed by Expert Assessor
Description: as for outcome 2
Time Frame: 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 460 | 460
percent of participants | 65 | 79

7. Secondary Outcome: Percentage of Participants Achieving Device Mastery at the End of Level 2 Out of a 6 Level Training Process at Week 8 as Assessed by Expert Assessor
Description: as for outcome 3
Time Frame: 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 460 | 460
percent of participants | 93 | 92

8. Secondary Outcome: Number of Participants Achieving Device Mastery at Levels 1-6 as Assessed by Expert Assessor
Description: Number of participants achieving mastery at each level in the 6 level training process at baseline visit as assessed by expert assessor
Time Frame: 0 weeks (Visit 1)
Measure: Number; unit: participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 516 | 516
participants
  Level 1: Intuitive Use | 20 | 113
  Level 2: Patient Information Leaflet | 142 | 186
  Level 3: Instructional Video | 176 | 87
  Level 4: Expert Tuition | 158 | 116
  Level 5: Repeat of Expert Tuition | 19 | 13
  Level 6: Second Repeat of Expert Tuition | 1 | 1

9. Secondary Outcome: Number of Participants Achieving Device Masteryin Levels 1-6 After 4 Weeks From Baseline Visit as Assessed by Expert Assessor
Description: Number of participants achieving mastery at each level in the 6 level training process after 4 weeks from baseline visit as assessed by expert assessor
Time Frame: 0 weeks (Visit 1)
Measure: Number; unit: participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 498 | 498
participants
  Level 1: Intuitive Use | 202 | 317
  Level 2: Patient Information Leaflet | 182 | 113
  Level 3: Instructional Video | 60 | 34
  Level 4: Expert Tuition | 47 | 31
  Level 5: Repeat of Expert Tuition | 7 | 3
  Level 6: Second Repeat of Expert Tuition | 0 | 0

10. Secondary Outcome: Number of Participants Achieving Device Mastery in Levels 1-6 After 8 Weeks From Baseline Visit as Assessed by Expert Assessor
Description: Number of participants achieving mastery at each level in the 6 level training process after 8 weeks from baseline visit as assessed by expert assessor
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 460 | 460
participants
  Level 1: Intuitive Use | 299 | 362
  Level 2: Patient Information Leaflet | 127 | 63
  Level 3: Instructional Video | 16 | 20
  Level 4: Expert Tuition | 14 | 19
  Level 5: Repeat of Expert Tuition | 0 | 0
  Level 6: Second Repeat of Expert Tuition | 0 | 0

11. Secondary Outcome: The Number of Levels Out of a 6 Level Training Process Required by Each Patient on Achieving Device Mastery as Assessed by Expert Assessor
Description: Number of levels required to achieve device mastery out of a 6 level training processrequired by each patient at each visit as assessed by expert assessor
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: levels
Groups:
- Budesonide/Formoterol (BF) Spiromax®: Training HCPs with a placebo comparator: Budesonide/Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: Budesonide/Formoterol (BF) Spiromax®: Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: SYMBICORT® Turbohaler: Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
- SYMBICORT Turbohaler®: Training HCPs with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: Budesonide/Formoterol (BF) Spiromax®: Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: SYMBICORT® Turbohaler: Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
Arm/Group | Budesonide/Formoterol (BF) Spiromax® | SYMBICORT Turbohaler®
Number analyzed (Participants) | 516 | 516
levels
  Visit 1 | 2.48 (1.15) | 3.03 (3.0)
  Visit 2 | 1.57 (0.91) | 1.94 (1.01)
  Visit 3 | 1.33 (0.73) | 1.45 (0.72)

12. Secondary Outcome: Number of Assessor-observed Errors Recalled During Baseline Visit by All Participants
Description: Quantity of errors made at each level recalled during baseline visit by all participants using an expert assessor
Time Frame: 0 weeks (Visit 1)
Measure: Number; unit: errors
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 516 | 516
errors | 2540 | 1447

13. Secondary Outcome: Number of Assessor-observed Errors Recalled at 4 Weeks After Baseline Visit by All Participants
Description: Quantity of errors made at each level recalled by expert assessors at 4 weeks after baseline visit by all participants
Time Frame: 4 weeks
Measure: Number; unit: errors
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 498 | 498
errors | 780 | 367

14. Secondary Outcome: Number of Assessor-observed Errors Recalled 8 Weeks After Baseline Visit by All Participants
Description: Quantity of errors made at each level recalled by expert assessors at 8 weeks after baseline visit by all participants
Time Frame: 8 weeks
Measure: Number; unit: errors
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Number analyzed (Participants) | 460 | 460
errors | 296 | 175

15. Secondary Outcome: Type of Participant Handling Errors Recalled by Expert Assessors at Baseline Visit by All Participants
Time Frame: 0 weeks (Visit 1)
Measure: Number; unit: errors
Arm/Group | Budesonide/Formoterol (BF) Spiromax® | SYMBICORT Turbohaler®
Number analyzed (Participants) | 516 | 516
errors
  Not holding device with mouthpiece cover at bottom | 62 | 0
  Device is not held upright (±90°) during dose prep | 318 | 0
  Device is not held upright (±45°) during dose prep | 0 | 614
  Not twisting the base until it clicks | 0 | 557
  Vigorous shaking before or after dose preparation | 78 | 29
  Exhales into the device before taking a dose | 61 | 101
  Inhalation is not as fast as possible from start | 613 | 581
  Does not remove cap | 0 | 6
  Inhaler not held upright (± 45°) until inhalation | 0 | 402
  Fails to seal lips around mouthpi | 131 | 157
  Puts fingers or mouth/face around air inlets | 105 | 93
  Does not open cap | 28 | 0
  A click is not heard when the cap is opened | 51 | 0

16. Secondary Outcome: Type of Participant Handling Errors by Expert Assessors 4 Weeks After Baseline Visit by All Participants
Time Frame: 4 weeks
Measure: Number; unit: errors
Arm/Group | Budesonide/Formoterol (BF) Spiromax® | SYMBICORT Turbohaler®
Number analyzed (Participants) | 498 | 498
errors
  Not holding device with mouthpiece cover at bottom | 6 | 0
  Device is not held upright (±90°) during dose prep | 106 | 0
  Device is not held upright (±45°) during dose prep | 0 | 184
  Not twisting the base until it clicks | 0 | 204
  Vigorous shaking before or after dose preparation | 19 | 8
  Exhales into the device before taking a dose | 23 | 36
  Inhalation is not as fast as possible from start | 148 | 166
  Does not remove cap | 0 | 0
  Inhaler not held upright (± 45°) until inhalation | 0 | 119
  Fails to seal lips around mouthpi | 15 | 20
  Puts fingers or mouth/face around air inlets | 0 | 43
  Does not open cap | 0 | 0
  A click is not heard when the cap is opened | 2 | 0

17. Secondary Outcome: Type of Participant Handling Errors Recalled by Expert Assessors 8 Weeks After Baseline Visit by All Participants
Time Frame: 8 weeks
Measure: Number; unit: errors
Arm/Group | Budesonide/Formoterol (BF) Spiromax® | SYMBICORT Turbohaler®
Number analyzed (Participants) | 460 | 460
errors
  Not holding device with mouthpiece cover at bottom | 3 | 0
  Device is not held upright (±90°) during dose prep | 34 | 0
  Device is not held upright (±45°) during dose prep | 0 | 70
  Not twisting the base until it clicks | 0 | 49
  Vigorous shaking before or after dose preparation | 6 | 2
  Exhales into the device before taking a dose | 12 | 19
  Inhalation is not as fast as possible from start | 71 | 82
  Does not remove cap | 0 | 0
  Inhaler not held upright (± 45°) until inhalation | 0 | 30
  Fails to seal lips around mouthpi | 5 | 5
  Puts fingers or mouth/face around air inlets | 41 | 39
  Does not open cap | 0 | 0
  A click is not heard when the cap is opened | 0 | 0

18. Secondary Outcome: Preference of Participant Device Questionnaire Assessed by PASAPQ Part II Q15 Score
Description: Device preference for either Spiromax or Turbohaler device at baseline assessed by PASAPQ Part II Q15 score
Time Frame: 0 weeks (Visit 1)
Measure: Number; unit: percent of participants
Groups:
- No Preference: HCPs indicated no preference of device during training with a placebo comparator: Budesonide/Formoterol (BF) Spiromax® device or placebo comparator: SYMBICORT® Turbohaler using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: Budesonide/Formoterol (BF) Spiromax®: Training with a placebo comparator: Budesonide Formoterol (BF) Spiromax® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
  Placebo Comparator: SYMBICORT® Turbohaler: Training with a placebo comparator: SYMBICORT Turbohaler® device using a 6-level system to examine the number of levels required to acquire mastery of device at baseline and maintenance and mastery at 4 and 8 weeks after initial training.
Arm/Group | Budesonide/Formoterol (BF) Spiromax® | SYMBICORT Turbohaler® | No Preference
Number analyzed (Participants) | 516 | 516 | 516
percent of participants | 74 | 16 | 10

19. Secondary Outcome: Preference of Device Questionnaire 4 Weeks After Baseline Visit Assessed by PASAPQ Part II Q15 Score
Description: Device preference for either Spiromax or Turbohaler device 4 weeks after baseline visit assessed by PASAPQ Part II Q15 score
Time Frame: 4 weeks
Measure: Number; unit: percent of participants
Arm/Group | Budesonide/Formoterol (BF) Spiromax® | SYMBICORT Turbohaler® | No Preference
Number analyzed (Participants) | 498 | 498 | 498
percent of participants | 74.5 | 15.5 | 10

20. Secondary Outcome: Preference of Device Questionnaire 8 Weeks After Baseline Visit Assessed by PASAPQ Part II Q15 Score
Description: Device preference for either Spiromax or Turbohaler device 8 weeks after baseline visit assessed by PASAPQ Part II Q15 score
Time Frame: 8 weeks
Measure: Number; unit: percent of participants
Arm/Group | Budesonide/Formoterol (BF) Spiromax® | SYMBICORT Turbohaler® | No Preference
Number analyzed (Participants) | 460 | 460 | 460
percent of participants | 79 | 14 | 7

ADVERSE EVENTS:
Time Frame: No adverse event data was collected.
Arm/Group | SYMBICORT Turbohaler® | Budesonide/Formoterol (BF) Spiromax®
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes